CLINICAL TRIAL: NCT00085774
Title: A Single-Dose Efficacy Comparison of Albuterol Hydrofluoroalkane (HFA) Breath-operated Inhaler (BOI) (Volare Easi-Breathe™) and Albuterol HFA Meter Dose Inhaler (MDI) (Volare™) in Adolescents and Adults With Exercise-Induced Bronchospasm
Brief Title: Comparison of Two Bronchodilator Inhalers in Adolescents and Adults With Exercise-Induced Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXR-302-4-167
Record Dates: First submitted 2004-06-14; First posted 2004-06-17 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Exercise-induced Bronchospasm
Keywords: albuterol; aerosol inhaler; metered-dose inhaler; breath-actuated inhaler; exercise-induced bronchospasm
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Albuterol HFA BOI (Experimental)
  Interventions: Drug: albuterol aerosol by HFA BOI
- Albuterol HFA MDI (Experimental)
  Interventions: Drug: albuterol aerosol by HFA MDI
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo aerosol by HFA

INTERVENTIONS:
Drug: albuterol aerosol by HFA MDI — albuterol HFA MDI 160 mcg
  Arms: Albuterol HFA MDI
Drug: albuterol aerosol by HFA BOI — albuterol HFA BOI 160 mcg
  Arms: Albuterol HFA BOI
Drug: placebo aerosol by HFA — placebo HFA
  Arms: Placebo

SUMMARY:
This study was designed to examine the effectiveness of two bronchodilator inhalers in patients who have exercise-induced asthma.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Male or non-pregnant, non-nursing females aged 12 40 years, inclusive, at the first screening visit
* Have exercise-induced bronchospasm (EIB), with or without asthma, as demonstrated by a ≥15% decrease in pre-challenge absolute FEV1 observed up to 60 minutes following an exercise challenge conducted at the first screening visit
* Predicted FEV1 ≥70% for age, height, gender, and, where applicable, race following an 8 hour period without [beta]2 agonist use
* Have no contraindications for exercising maximally
* Ability to perform spirometry reproducibly (i.e., the difference between the two highest FEV1 values out of a minimum of three and a maximum of eight values obtained at the first screening visit must not exceed 0.2 L)
* Ability to self-perform PEF (peak expiratory flow) determinations with a handheld peak flow meter
* Can tolerate withdrawal of applicable medications for qualification at both screening visits
* Normal chest X ray, or, if abnormal, is consistent with asthma and shows no evidence of other active disease
* Otherwise healthy individuals with clinically acceptable medical history, physical examination, vital signs, and 12 lead ECG (electrocardiogram; with 30 second Lead II rhythm strip)
* Body mass index (BMI) of 19 29 kg/m2 (BMI = weight [kg] / height2 [m])
* Non-smokers for at least one year prior to the first screening visit and have maximum smoking histories of ten-pack years (i.e., equivalent to 20 cigarettes per day for 10 years).

Exclusion Criteria:

* Allergy or sensitivity to albuterol or to other components of the formulations used in the drug
* Exposure to investigational drugs within 30 days prior to the first screening visit
* Require continuous treatment with [beta] blockers (administered by any route), MAO (monoamine oxidase) inhibitors, tricyclic antidepressants, cromones (by any route), antileukotrienes, and/or systemic corticosteroids
* Treated with oral or injectable corticosteroids within the 12 weeks prior to the first screening visit
* The prescribed dose regimen of any required inhaled corticosteroids has not been stable for at least four weeks prior to the first screening visit NOTE: Patients requiring subsequent dosage adjustment of these drug products must be discontinued from the study.
* Inability to tolerate or unwillingness to comply with required washout periods for all applicable medications and xanthine-containing foods and beverages prior to the screening visit
* Treatment in an emergency room for asthmatic symptoms or hospitalization for asthmatic symptoms within twelve months prior to the first screening visit
* Experienced an upper respiratory tract infection and/or sinusitis associated with exacerbation of asthmatic symptoms not requiring emergency room treatment and/or hospitalization and/or treatment with oral or injected corticosteroids that has not resolved within four weeks prior to the screening visit
* History and/or presence of any clinically-significant acute or chronic disease, including but not limited to bronchitis, emphysema, active tuberculosis, bronchiectasis, cystic fibrosis, clinically significant cardiovascular disease (including cardiac arrhythmias and uncontrolled hypertension), clinically significant hepatic, renal, or endocrine dysfunction, stroke, uncontrolled diabetes, hyperthyroidism, convulsive disorders, and neoplastic disease other than basal cell carcinoma of the skin
* Known or suspected substance abuse (e.g., alcohol, marijuana, etc.) and/or presence of any other medical or psychological conditions that in the investigator's opinion should preclude study enrollment.
* Are employees of this study site or have a family member associated with the conduct of this study at this site
* Previous enrollment in an IVAX Research-sponsored Albuterol HFA aerosol asthma study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2004-09-30 (Actual); Study Completion 2004-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was mean maximum % change in the baseline absolute forced expiratory volume in 1 second (FEV1) value observed up to 1 hour post-challenge. | Three doses 2-7 days apart

SECONDARY OUTCOMES:
Mean maximum percent change in the baseline percent predicted FEV1 value observed up to one hour post-challenge | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean maximum absolute change in the baseline absolute FEV1 value observed up to one hour post-challenge | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean percent change in the baseline absolute FEV1 value at each post-challenge time point | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean absolute change in the baseline absolute FEV1 value at each post-challenge time point | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean percent change in the baseline percent-predicted FEV1 value at each post-challenge time point | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean largest negative (or mean smallest positive) percent change in the baseline absolute FEV1 value observed up to one hour post-challenge | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Mean largest negative (or mean smallest positive) percent change in the average test-day pre-dose baseline percent predicted FEV1 value observed up to one hour post-challenge | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Time to recovery (in minutes) measured from time of completion of exercise challenge to time FEV1 returns to 10% or less of baseline value during the recovery phase | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Total changes in FEV1 expressed as the baseline-adjusted area-under-the-effect curve of the percent-predicted FEV1 versus time over 60 minutes (AUEC0 60) | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes
Percentage of patients who are "protected" (maximum percent decrease in the baseline absolute FEV1 <10%), "partially protected" (10 20%), and "unprotected" (>20%). | exercise challenge 30 minutes after dosing and assessments over 60 +/- 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David S Pearlman, MD, Principal Investigator — Colorado Allergy and Asthma Centers, PC
Locations (3):
- United States (3):
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Colorado Allergy and Asthma Centers, PC, Englewood, Colorado
  - Colorado Allergy and Asthma Centers, PC, Lakewood, Colorado